CLINICAL TRIAL: NCT06189495
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetic Profile of Genakumab Injection in Patients With Connective Tissue Disease-associated Interstitial Lung Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GenSci048-204
Record Dates: First submitted 2023-11-13; First posted 2024-01-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Systemic Sclerosis Associated Interstitial Lung Disease; Rheumatoid Arthritis Associated Interstitial Lung Disease (RA-ILD); Systemic Sclerosis Associated Interstitial Lung Disease (SSc-ILD)
Keywords: connective tissue disease-associated interstitial lung disease; Rheumatoid Arthritis associated Interstitial Lung Disease (RA-ILD); Systemic Sclerosis associated Interstitial Lung Disease (SSc-ILD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GenSci048 (Experimental): 1. Dosage: 300 mg.2. Duration of administration: All subjects received one dose of Genakumab injection every 4 weeks according to their group.The dose was injected subcutaneously.3. Course of administration: Phase I subjects were treated with Genakumab injection until the end of the study or the occurrence of the drug.Tolerable toxicity or investigator-assessed efficacy (whichever occurs first); The phase 2 randomized double-blind treatment period was 24 weeks, with a total of 6 administration times. After the randomized double-blind treatment period, an open-label treatment period was entered, and all subjects will receive Genakumab injection 300 mg Q4W until the end of the study or the occurrence of intolerable toxicity or poor efficacy assessed by the investigators (whichever occurs first).4. Administration method: subcutaneous injection; The injection site is the abdomen (3 cm away from the navel
  Interventions: Drug: GenSci048
- GenSci048 placebo (Placebo Comparator): .1. Dosage: 300 mg.2. Duration of administration: All subjects received one dose of placebo every 4 weeks according to their group The dose was injected subcutaneously.3. Course of administration: Phase I subjects were treated with placebo until the end of the study or the occurrence of the drug.Tolerable toxicity or investigator-assessed efficacy (whichever occurs first); The phase 2 randomized double-blind treatment period was 24 weeks, with a total of 6 administration times. After the randomized double-blind treatment period, an open-label treatment period was entered, and all subjects will receive placebo 300 mg Q4W until the end of the study or the occurrence of intolerable toxicity or poor efficacy assessed by the investigators (whichever occurs first).
  4. Administration method: subcutaneous injection; The injection site is the abdomen (3 cm away from the navel)
  Interventions: Drug: GenSci048 placebo

INTERVENTIONS:
Drug: GenSci048 — 1. Dosage: 300 mg.2. Duration of administration: All subjects received one dose of Genakumab injection every 4 weeks according to their group.The dose was injected subcutaneously.3. Course of administration: Phase I subjects were treated with Genakumab injection until the end of the study or the occurrence of the drug.Tolerable toxicity or investigator-assessed efficacy (whichever occurs first); The phase 2 randomized double-blind treatment period was 24 weeks, with a total of 6 administration times. After the randomized double-blind treatment period, an open-label treatment period was entered, and all subjects will receive Genakumab injection 300 mg Q4W until the end of the study or the occurrence of intolerable toxicity or poor efficacy assessed by the investigators (whichever occurs first).4. Administration method: subcutaneous injection; The injection site is the abdomen (3 cm away from the navel
  Arms: GenSci048
Drug: GenSci048 placebo — 1. Dosage: 300 mg.2. Duration of administration: All subjects received one dose of placebo every 4 weeks according to their group The dose was injected subcutaneously.3. Course of administration: Phase I subjects were treated with placebo until the end of the study or the occurrence of the drug.Tolerable toxicity or investigator-assessed efficacy (whichever occurs first); The phase 2 randomized double-blind treatment period was 24 weeks, with a total of 6 administration times. After the randomized double-blind treatment period, an open-label treatment period was entered, and all subjects will receive placebo 300 mg Q4W until the end of the study or the occurrence of intolerable toxicity or poor efficacy assessed by the investigators (whichever occurs first).
  4. Administration method: subcutaneous injection; The injection site is the abdomen (3 cm away from the navel)
  Arms: GenSci048 placebo

SUMMARY:
This study was conducted in a randomized, double-blind, placebo-controlled design to evaluate the efficacy and safety of Genakumab injection in the treatment of CTD-ILD including Rheumatoid Arthritis associated Interstitial Lung Disease (RA-ILD) and Systemic Sclerosis associated Interstitial Lung Disease (SSc-ILD)

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily sign informed consent and can complete the experiment according to the plan;
2. Age 18-75 years old (including upper and lower limits), both male and female;
3. Rheumatoid arthritis (RA) diagnosed according to the 2010 American College of Rheumatology (ACR)/European League against Rheumatism (EULAR) classification, or Systemic sclerosis (SSc) according to the 2013 ACR/EULAR classification;
4. Interstitial lung disease (ILD) was confirmed by HRCT within 12 months before screening.
5. FVC≥ 40% of the expected value during the screening period;
6. DLCO (using hemoglobin correction) ≥ 40% of the expected value during the screening period;
7. Patients may receive 1 immunosuppressant and must maintain a stable dose for 3 months prior to the first dose and agree to maintain a stable dose for at least 6 months after the first dose;
8. Subjects of childbearing age who do not plan to become pregnant or donate sperm/eggs and agree to use reliable contraception during the period of participation in this trial and within 6 months after the last dosing.

Exclusion Criteria:

1. Allergic to experimental drugs or biological agents; People who have previously known other severe allergic reactions;
2. Airway obstruction (FEV1/FVC<0.7 before bronchodilator use) or other lung abnormalities deemed clinically significant by the investigator or a history of asthma;
3. Those who have received any of the following drugs or treatments :

   1. Receiving prednisone >15mg/ day or equivalent dose of glucocorticoid within 2 weeks prior to randomization;
   2. Receive azathioprine, colchicine, D-penicillamine, sulfasalazine within 8 weeks before randomization;
   3. received rituximab, tolizumab, nidanib, pirfenidone and other treatments within 6 months before randomization; Abacil, TNF inhibitors and other biologic agents were received within 3 months before randomization; Tofaciib, tacrolimus, cyclosporin A, and potassium para-aminobenzoate were used 30 days or 5 half-lives prior to screening, whichever was older.
4. Combined with other rheumatic diseases, such as idiopathic inflammatory myopathy, systemic lupus erythematosus, Sjogren's syndrome, mixed connective tissue disease, systemic vasculitis;
5. Significant pulmonary hypertension, meeting one of the following conditions:

   1. Previous clinical or echocardiographic evidence of significant right heart failure;
   2. Right cardiac catheterization showed cardiac index ≤ 2 l/min/m2;
   3. Pulmonary hypertension requiring extraenteral treatment with eprostol/traprostacycline;
6. There are active bleeding diseases of internal organs, or have a serious bleeding tendency (such as hemophilia, etc.), or are undergoing anticoagulant treatment;
7. There are infections requiring systemic drug control within 7 days prior to screening; Diagnosed with active tuberculosis infection;
8. Have received live or attenuated vaccine within 3 months prior to screening, or plan to receive live or attenuated vaccine during the study period; Vaccination against COVID-19 within 2 weeks prior to screening;
9. Previous stem cell therapy or any type of bone marrow transplant; Previous solid organ transplants; Long-term systemic use of glucocorticoids for other diseases;
10. There is a history of serious immunodeficiency, or other acquired or congenital immunodeficiency diseases;
11. History of malignant tumor within 5 years before screening;
12. Recipients of kidney dialysis;
13. Presence of the following clinically significant heart diseases:

    1. A history of chronic congestive heart failure, NYHA level IV; History of cardiac ejection fraction (EF) < 30% by echocardiography;
    2. Myocardial infarction, acute coronary syndrome, viral myocarditis, and pulmonary embolism occurred within 3 months; Coronary revascularization was performed within 6 months.
    3. There are severe arrhythmias that require Class Ia or III antiarrhythmic drugs; Arrhythmias with diseased sinus syndrome, grade II type II or grade III atrioventricular block, and no pacemaker implanted;
    4. During the screening period, electrocardiogram indicated QTcF interval ≥ 480 ms (according to Fridericia correction formula, where QTcF=QT/RR^0.33), or a history of prolonged QTc interval;
14. There are the following abnormalities in the laboratory test values during the screening period:

    1. White blood cell count <3×109/L, neutrophil count <1.5×109/L;
    2. PLT<75×109/L;
    3. Total bilirubin >1.5×ULN, alanine aminotransferase (ALT) >3×ULN, aspartate aminotransferase (AST) >3×ULN;
    4. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2;
15. History or current positive results of serum virology tests:

    1. hepatitis B surface antigen positive, or hepatitis B core antibody positive and HBV-DNA higher than the detection limit;
    2. Hepatitis C virus (HCV) antibody positive;
    3. Positive for human immunodeficiency virus (HIV) antibodies;
    4. Those who are positive for treponema pallidum antibodies and need treatment for syphilis infection.
16. Received treatment with any investigational drug or medical device in a clinical trial within 3 months prior to screening;
17. Pregnancy test positive during screening period; Lactating women;
18. The investigator assessed those who had other factors that made them unsuitable for participation in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Lung function assessment:Subjects' lung function was assessed by FVC . | FVC will be evaluated simultaneously during the screening period, 4 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks, and once every 24 weeks thereafter, From baseline up to 2 years
Lung function assessment:Subjects' lung function was assessed by DLCO. | DLCO will be evaluated simultaneously during the screening period, 4 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks, and once every 24 weeks thereafter, From baseline up to 2 years，early withdrawal/termination of treatment, and when the investigator deems
tLung function assessment:Visual simulation score was used to evaluate Physician's Global Asseessment（PGA） | "Lung function assessment:The PGA is evaluated during the screening period and once every 12 weeks .From baseline up to 2 years.
Safety evaluation indicator：Adverse Events | From baseline up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: qibing xie, Doctor of Medicine(M.D.), Study Chair — West China Hospital
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan